CLINICAL TRIAL: NCT00352144
Title: A Six-Month, Chronic Efficacy and Safety Study of Eszopiclone in Adult Subjects With Primary Insomnia: A Randomized Double-Blind, Placebo-Controlled Study
Brief Title: 6-Month Chronic Efficacy & Safety Study of Eszopiclone in Adult Subjects With Primary Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-050
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): eszopiclone 3 mg tablet
  Interventions: Drug: Eszopiclone
- 2 (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3 mg
  Other Names: Lunesta; S-Zopiclone
  Arms: 1
Drug: Placebo — Placebo tablet
  Arms: 2

SUMMARY:
To evaluate the long-term efficacy of eszopiclone administered for up to 6 months in subjects with primary insomnia on subjective sleep measures, compared to placebo.

DETAILED DESCRIPTION:
This is a double blind, randomized (2:1; eszopiclone : placebo), placebo-controlled, multicenter, study of eszopiclone in subjects with primary insomnia. The study will involve up to 9 visits and subject participation will be approximately 224 days. After meeting all screening criteria, subjects will be randomized to either eszopiclone 3 mg QD or placebo. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Subject meets DSM-IV criteria for primary insomnia and reports sleeping no more than 6.5 hours per night and/or taking more than 30 minutes each night to fall asleep for at least one month prior to screening.
* Male and female subjects must be between 21 and 64 years of age, inclusive, at the time of consent.
* Female subjects of childbearing potential must sign the Women of Childbearing Potential Addendum to the informed consent form. Females considered not of childbearing potential must be surgically sterile or greater than one-year post menopausal, defined as a complete cessation of menstruation for at least one year.
* Subject must be in general good health, based on screening physical examination (including brief neurological examination), medical history, 12-lead ECG, and clinical laboratory values (hematology, serum chemistry and urinalysis).

Exclusion Criteria

* Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, respiratory, hepatic, or renal systems.
* Subject has a history of cancer within the past 5 years, or current malignancy except for non melanomatous skin cancer.
* Subject has a psychiatric diagnosis with psychosis, dementia or delirium. Subjects with Sexual and Gender Identity Disorders or other non-psychotic disorders will be considered on a case-by-case basis.
* Subject has one of the following Personality Disorders: schizotypal, schizoid, or borderline personality disorder.
* Subject has difficulties in sleep initiation or maintenance associated with known medical diagnosis (e.g. sleep apnea, restless leg syndrome (RLS), or periodic leg movement syndrome (PLMS), or has any condition that has or may affect sleep (e.g., chronic pain, BPH, etc.).
* Subject has participated in a previous eszopiclone clinical trial.
* Subject has a known sensitivity to racemic zopiclone, any benzodiazepine, any sedative hypnotic, any substance that is contained in the formulation, or has been hospitalized for any allergic conditions (e.g. recurrent dermatitis, drug hypersensitivity, drug allergy, etc.).
* Subject has history of substance abuse in the past 10 years or substance dependence at any time or positive urine drug test at screening .
* Subject tests positive at screening for hepatitis B surface antigen, hepatitis C antibody or has a history of a positive result.
* Subject is known to be seropositive for HIV.
* Female subjects who are pregnant, lactating or within 6 months post partum.
* Subject self-reports consumption of more than two alcoholic beverages daily, 14 or more alcoholic beverages weekly, or five or more alcoholic beverages on any given day.
* Subject has taken any psychotropic medications or other medications known to affect sleep within the 3 days prior to screening visit or is anticipated to need any of these types of medications during double-blind treatment .
* Subject has participated in any investigational study within 30 days prior to screening.
* Subject has taken herbal supplements, purported to have central nervous system effects,(tablets, powders, extracts or tinctures) or combination products with herbs or melatonin within 14 days prior to screening or St. John's Wort within 30 days prior to screening.
* Subject is a rotating or third/night shift worker.
* Subject is a staff member or relative of a staff member.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 830 (Actual)
Dates: Start 2003-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Average of Subjective Sleep Latency | Days -14, 1, 30, 60, 90, 120, 150, 180

SECONDARY OUTCOMES:
Average of Total Sleep Time (TST) and Wake Time After Sleep Onset (WASO) | Days -14, 1, 30, 60, 90, 120, 150, 180
SF-36 | Days 1, 30, 90, 180
Work Limitations Questionnaire (WLQ) | Days 1, 30, 90, 180
Insomnia Severity Index (ISI) | Days 1, 30, 90, 180
Fatigue Severity Scale (FSS) | Days 1, 30, 90, 180
Epworth Sleepiness Scale (ESS) | Days 1, 30, 60, 90, 120, 150, 180
Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ) | Day 180
Healthcare Utilization Questionnaire (HUQ) | Days 1, 30, 60, 90, 120, 150, 180

CONTACTS AND LOCATIONS:
Locations (58):
- United States (58):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Anaheim, California
  - Irvine, California
  - Oakland, California
  - Redlands, California
  - San Diego, California
  - Aurora, Colorado
  - Denver, Colorado
  - Longmont, Colorado
  - Pueblo, Colorado
  - Clearwater, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Naples, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Blairsville, Georgia
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Northbrook, Illinois
  - Evansville, Indiana
  - Olathe, Kansas
  - Prairie Village, Kansas
  - Chevy Chase, Maryland
  - Frederick, Maryland
  - Newton, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Hamilton, New Jersey
  - New York, New York
  - Cary, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Jackson, Texas
  - Lubbock, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Brown Deer, Wisconsin
  - Madison, Wisconsin